CLINICAL TRIAL: NCT00073268
Title: Prevention of Type 2 Diabetes Mellitus in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 14239 (completed)
Record Dates: First submitted 2003-11-18; First posted 2003-11-19 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; adolescent
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
This is a pilot study to examine the short-term effects of supervised exercise on metabolic risk factors for type 2 diabetes mellitus in children from a population that is at high risk for this disease. We hypothesize that exercise will significantly improve insulin sensitivity in all children, especially in children who are already insulin resistant, thereby lowering the risk that they will go on to develop type 2 diabetes mellitus. The specific hypotheses being tested are:

1. Insulin resistance will be most evident in overweight children while an impaired ability of the pancreas to release insulin will be most evident in children with a family history of type 2 diabetes mellitus.
2. Exercise will significantly improve insulin resistance (as measured by the fasting glucose/insulin ratio) with little or no effect on insulin secretory capacity (as measured by circulating insulin concentration at 1, 3, and 5 minutes following an intravenous glucose load) in children.
3. Participation in a school-based health, nutrition, and exercise education program will have long-term beneficial effects on health-related behaviors and on insulin resistance.

ELIGIBILITY:
Early adolescent

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2002-12; Study Completion 2007-06

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Russ Berrie Pavilion, New York, New York
  - New York Presbyterian Hospital, New York, New York